CLINICAL TRIAL: NCT03770520
Title: The Clinical Effect of QFR-guided Coronary Artery Bypass Grafting: a Randomized Controlled Trial
Brief Title: Graft Patency of QFR-guided Versus Angio-guided Coronary Artery Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Dong Ran, Direcotr,chief of ward No.11, Department of cardiac surgery, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z171100001017059
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: Quantitative Flow Ratio; Coronary Artery Bypass Grafting; Graft patency
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: QFR will be masked to care providers and participants, and open to investigators, the allocation will be based on QFR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QFR-guided (Experimental): This group will be performed a CABG surgery based on CAG and QFR, whether graft the moderate stenosis vessels will be based on the result of QFR.
  Interventions: Procedure: QFR-guided CABG
- Angio-guided (Active Comparator): This group will be performed a CABG surgery only based on CAG, the final surgery strategy will be decided after the discussion of heart team.
  Interventions: Procedure: Angio-guided CABG

INTERVENTIONS:
Procedure: QFR-guided CABG — CABG surgery based on CAG and QFR
  Arms: QFR-guided
Procedure: Angio-guided CABG — CABG surgery based on heart team discussion of CAG
  Arms: Angio-guided

SUMMARY:
Coronary artery bypass grafting(CABG) is the golden standard for severe coronary artery disease(CAD), the current surgery strategy is mainly based on coronary angiography(CAG), but many trials of PCI have shown that visually stenosis in CAG may not have functional significance. The aim of this study is to investigate if the Quantitative Flow Ratio (QFR) can be adopted in CABG and achieve a better graft patency.

DETAILED DESCRIPTION:
CABG is the major treatment of three vessels or left main disease. CAG is the main basis on choosing the vessels to graft, however, some of the grafts occluded shortly after surgery due to competitive flow, these vessels may not be significantly stenosis in functional assessment such as Fractional Flow Reserve (FFR). Quantitative Flow Ratio (QFR) is a novel method for evaluating the functional significance of coronary stenosis. Comparing to FFR, there is no need for pressure wire or ATP when performing QFR. This study plan to investigate the clinical effect of QFR in CABG, all patients included will be allocated 1:1 into two groups: QFR-guided and Angio-guided, QFR-guided group will be performed a CABG based on the result of QFR, the other group will be based on heart team discussion of CAG, CTA will be adopted to evaluate the 1 year graft patency.

ELIGIBILITY:
Inclusion Criteria:

* patients with evidence of angina pectoris
* left main or three vessels disease, have the indication for CABG after discussion of the heart team
* at least one main vessels stenosis on 40%-70%

Exclusion Criteria:

* former cardiac surgery patients
* need to perform other cardiac or major surgery( i.e. valve surgery, carotid endarterectomy
* emergent CABG
* acute myocardial infarction time less than 7 days
* life expectancy less than 3 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
The rate of graft patency | 12 months
  graft patency will be evaluated by CTA, 2 doctors will be invited to read the CT and draw their own conclusion without knowing the other result

SECONDARY OUTCOMES:
Major adverse cardiovascular event(MACE) | 12 months
  The rate of deaths due to cardiovascular events, myocardial infarction and second revascularization
The rate of angina relief | 12 months
  whether angina is relieved will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Ran Dong, MD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided